CLINICAL TRIAL: NCT01128790
Title: Effect of Remote Ischemic Preconditioning on Exercise Capacity in Patients With Heart Failure: A Double Blind Randomized Control Trial
Brief Title: Pilot Study of Remote Ischemic Preconditioning in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-0550-BE
Record Dates: First submitted 2009-12-17; First posted 2010-05-24 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Heart Failure; Left Ventricular Dysfunction
Keywords: exercise; remote ischemic preconditioning; heart failure; left ventricular dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- remote ischemic preconditioning (Experimental): 4 cycles of 5 mins upper limb ischemia induced by blood pressure cuff inflation 20mmHg above systolic blood pressure
  Interventions: Other: Remote ischemic preconditioning
- Sham control (Sham Comparator): 4 x 5 mins of upper limb blood pressure cuff inflation to 10mmHg (non-occlusive)
  Interventions: Other: Sham Control

INTERVENTIONS:
Other: Remote ischemic preconditioning — 4 cycles x 5 mins upper limb blood pressure cuff inflation 20mmHg above systolic blood pressure
  Arms: remote ischemic preconditioning
Other: Sham Control — 4 cycles x 5mins blood pressure cuff inflation to 10mmHg
  Arms: Sham control

SUMMARY:
The purpose of this study is to determine the effect of remote ischemic preconditioning on exercise capacity in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* LV ejection fraction <40%
* NYHA functional class II-IV
* Non ischemic cardiomyopathy
* Stable

Exclusion Criteria:

* recent cardiovascular hospitalization (within last 4 weeks)
* ischemic cardiomyopathy
* diabetes mellitus
* peripheral neuropathy
* ventricular assist device
* contraindications to exercise stress testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Exercise performance - VO2, exercise time, exercise workload, anaerobic threshold | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Brindle HE, Tetsa-Tata D, Edwards T, Choi EM, Kasonia K, Aboubacar S, Mambula G, Kavunga-Membo H, Grais R, Johnson J, Bausch DG, Muyembe-Tamfum JJ, Ama IS, Lees S, Watson-Jones D, Camacho A, Roberts CH. Using an analogue-digital hybrid clinical data management platform during a two-dose preventive Ebola virus vaccine trial in Goma, the Democratic Republic of the Congo. PLOS Glob Public Health. 2025 May 2;5(5):e0004487. doi: 10.1371/journal.pgph.0004487. eCollection 2025. PMID 40315243
- [Derived] McDonald MA, Braga JR, Li J, Manlhiot C, Ross HJ, Redington AN. A randomized pilot trial of remote ischemic preconditioning in heart failure with reduced ejection fraction. PLoS One. 2014 Sep 2;9(9):e105361. doi: 10.1371/journal.pone.0105361. eCollection 2014. PMID 25181050